CLINICAL TRIAL: NCT00853996
Title: Phase II Study of Acolbifene in Pre-Menopausal Women at High Risk for Breast Cancer
Brief Title: Acolbifene in Preventing Cancer in Premenopausal Women at High Risk of Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carol Fabian, MD, Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2009-01116; 10588 (Other: KUMC IRB); NCT00855751 (Registry Identifier: Clinical Trials.gov (obselete)); UW105-6-01 (Other: University of Wisconsin); N01CN35153 (NIH); NCT00855751 (obsolete NCT alias)
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prevention (acolbifene hydrochloride) (Experimental): Patients receive oral acolbifene hydrochloride once daily for 6 months in the absence of unacceptable toxicity.
  Interventions: Drug: acolbifene hydrochloride

INTERVENTIONS:
Drug: acolbifene hydrochloride — Given orally
  Other Names: EM-652.HCL; SCH 57068.HCl

SUMMARY:
This phase II trial is studying how well acolbifene works in preventing cancer in premenopausal women at high risk of breast cancer. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of acolbifene may stop cancer from growing or coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of six months of acolbifene 20 mg/day on Ki-67 in high risk premenopausal women with baseline hyperplasia +/- atypia and Ki-67 positivity of >= 2%..

SECONDARY OBJECTIVES:

I. To determine the effect of six months of acolbifene 20 mg/day on mammographic breast density in high risk premenopausal women.

II. To determine the effect of six months of acolbifene 20 mg/day on serum levels of follicular phase bioavailable estradiol, and luteal phase progesterone, testosterone, and fasting IGF-1/IGFBP-3.

III. To determine the effect of six months of acolbifene 20 mg/day on epithelial cell cytomorphology and molecular markers such as ER, PgR, and pS2.

IV. To determine the effect of six months of acolbifene on markers of cardiovascular risk (C-reactive protein, functional AntiThrombin III, and fasting lipid profile) and bone turnover markers associated with bone mineral density gain or loss (serum osteocalcin and N-telopeptide crosslinks).

V. To assess any increase in reported hot flashes, menstrual cycle irregularities, pelvic pain, musculoskeletal complaints, and fatigue from baseline.

OUTLINE:

Patients receive oral acolbifene hydrochloride once daily for 6 months in the absence of unacceptable toxicity.

Patients undergo symptom assessment (hot flashes, menstrual abnormalities, pelvic pain, muscle and joint pain, and fatigue) at baseline, 6-8 weeks, monthly for 6 months, and then at 2 weeks after completion of study treatment.

Patients undergo random periareolar fine needle aspiration between days 1-10 of menstrual cycle at baseline and at 6 months. Patients also undergo blood sample collection between days 1-10 and days 20-24 of menstrual cycle at baseline and at 6 months. Samples taken between days 1-10 of menstrual cycle are analyzed for Ki-67 expression, cytomorphology, molecular markers (estrogen receptor, progesterone receptor, and pS2 expression), and bioavailable estradiol levels. Samples taken between days 20-24 of menstrual cycle are analyzed for progesterone, testosterone, IGF-1, IGFBP-3, lipid profile, bone-turnover markers (osteocalcin and N-telopeptide crosslinks), C-reactive protein, and functional antithrombin III.

After completion of study treatment, patients are followed at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Gail risk >= 1.7% and/or relative risk >= 3 times that for 5-year age group
* Premenopausal
* More than 6 months since initiating or discontinuing oral contraceptives
* At increased risk for breast cancer, as indicated by >= 1 of the following risk factors:
* BRCA1/2 mutation characterized as deleterious or of uncertain significance
* Prior atypical ductal hyperplasia, ductal carcinoma in situ, or lobular carcinoma in situ
* Prior random periareolar fine needle aspiration (RPFNA) showing atypical hyperplasia
* Family history consistent with hereditary breast cancer, as indicated by 1 of the following criteria:

  * >= 4 relatives with breast cancer
  * >= 2 relatives diagnosed with breast cancer at ≤ 50 years of age
  * Breast and ovarian cancer diagnosed in same relative
* No suspicion for breast cancer on baseline mammogram performed between days 1-10 of menstrual cycle within 3 months prior to screening baseline RPFNA
* Exhibits hyperplasia with or without atypia (Masood score >= 14) with >= 500 cells AND Ki-67 positivity >= 2% by RPFNA performed within 6 months prior to initiation of study drug
* Estimated visual mammographic breast density category >= 5% on mammogram performed within 6 months prior to initiation of study drug
* Has regular menstrual cycles (between 21 and 35 days) unless using extended regimen oral contraceptives or a contraceptive device (e.g., Mirena IUD) Values for metabolic profile and blood count within normal limits
* Absolute granulocyte count > 1,000/mm^3
* Platelets > 100,000/mm^3
* Hemoglobin > 10 g/dL
* Bilirubin < 2.0 mg/dL
* AST < 2 times upper limit of normal (ULN)
* Albumin > 3.0 g/dL
* Creatinine < 1.5 mg/dL
* Alkaline phosphatase < 2 times ULN
* Concurrent hormonal contraceptives allowed provided patient remains on the same hormonal regimen from 3 months prior to baseline aspiration until the completion of study treatment
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Willing to ingest recommended dose of calcium and vitamin D for premenopausal bone health (1,200 mg calcium and 800 IU vitamin D daily)
* Negative pregnancy test prior to receiving study agent

Exclusion Criteria

* pregnant or nursing
* nursing within the past 6 months
* Known osteoporosis or severe osteopenia (T-score -2 or worse by DEXA)
* History of symptomatic endometriosis with pelvic pain, poorly controlled migraines, or hot flashes
* History of deep venous thrombosis
* History of allergic reactions attributed to compounds of similar chemical or biological composition to the study agent
* Other condition or concurrent illness that, in the opinion of the investigator, would make the patient a poor candidate for RPFNA
* Less than 1 year since prior use of aromatase inhibitors (e.g., anastrozole, exemestane, or letrozole) or selective estrogen receptor modulators (e.g., tamoxifen citrate, raloxifene, or arzoxifene hydrochloride)
* Other concurrent chemopreventive agents
* Concurrent anticoagulants
* Other concurrent investigational agents
* Bilateral breast implants

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Fabian, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared; only summary assessments.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevention (Acolbifene Hydrochloride)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (Acolbifene Hydrochloride)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Height [Mean (Standard Deviation); unit: inches] | 65 (2)
Weight [Mean (Standard Deviation); unit: pounds] | 155 (29)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.8 (4.8)
5-Year Gail Risk [Mean (Standard Deviation); unit: Percent risk of developing breast cancer] — Projected risk of a women developing breast cancer within the next 5 years, as calculated using the Gail Risk Model.
  Percent risk of developing breast cancer | 3.6 (4.4)
Age First Live Birth [Mean (Standard Deviation); unit: years] | 28 (4)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Percentage of Breast Epithelial Cells Expressing Ki-67, From Baseline to 6 Months
Description: Change in proliferation as measured by Ki-67 immunocytochemical expression in breast epithelial cells obtained by random periareolar fine needle aspiration at baseline and at 6 months.
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: percentage of positive cells
Arm/Group | Prevention (Acolbifene Hydrochloride)
Number analyzed (Participants) | 25
percentage of positive cells | -3.0 [-20.2 to 2.8]
Statistical Analysis 1: Comparison: Prevention (Acolbifene Hydrochloride); Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons since this was primary endpoint. A priori threshold for statistical significance was set at <0.05

2. Secondary Outcome: Change in Mammographic Breast Density
Description: Change in mammographic density from baseline to 6 months, The Percent Breast Density is estimated using the Cumulus computer-assisted program to define a region that is at greater density than the remainder of the breast.
Time Frame: Baseline to 6 months
Population: One subject was without a digital file due to technical reasons. Thus, only 24 subjects were evaluated.
Measure: Median (Inter-Quartile Range); unit: percentage of area at increased density
Arm/Group | Prevention (Acolbifene Hydrochloride)
Number analyzed (Participants) | 24
percentage of area at increased density | -3.9 [-31.4 to 16.2]
Statistical Analysis 1: Comparison: Prevention (Acolbifene Hydrochloride); Test type: Other; p = 0.067, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. A priori threshold for statistical significance was set at <0.05

3. Secondary Outcome: Change in Serum Estradiol Concentration
Description: Change in serum concentration of estradiol from baseline to 6 months
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Prevention (Acolbifene Hydrochloride)
Number analyzed (Participants) | 25
ng/ml | 64.6 (138)
Statistical Analysis 1: Comparison: Prevention (Acolbifene Hydrochloride); Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. A priori threshold for statistical significance was set at <0.05

4. Secondary Outcome: Change in Serum Concentration of Bioavailable Estradiol
Description: Change in serum concentration of bioavailable estradiol (adjusted for concentration of Sex Hormone Binding Globulin), from baseline to 6 months
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: pM
Arm/Group | Prevention (Acolbifene Hydrochloride)
Number analyzed (Participants) | 25
pM | 2.6 (7.0)
Statistical Analysis 1: Comparison: Prevention (Acolbifene Hydrochloride); Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. A priori threshold for statistical significance was set at <0.05

5. Secondary Outcome: Change in Serum Concentration of Testosterone
Description: Change in serum concentration of Testosterone from baseline to 6 months
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Prevention (Acolbifene Hydrochloride)
Number analyzed (Participants) | 25
ng/ml | 0.22 (0.48)
Statistical Analysis 1: Comparison: Prevention (Acolbifene Hydrochloride); Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. A priori threshold for statistical significance set at 0.05

6. Secondary Outcome: Reports of Hot Flashes as Assessed by the Loprinzi Hot Flash Scoring System
Description: Problems with hot flashes were assessed by average number per day and intensity.
Time Frame: Baseline to up to 2 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Acolbifene Hydrochloride)
Number analyzed (Participants) | 25
Participants
  Increase in hot flash frequency and/or severity | 6
  No change in hot flash frequency and/or severity | 14
  Decrease in hot flash frequency and/or severity | 5

7. Secondary Outcome: Reports of Muscle/Joint Complaints as Assessed by the Validated HAQ II Questionnaire
Description: The Health Assessment Questionnaire II (HAQ-II) measures interference in daily activities from arthralgias and joint pain. Range 0 - 4. A higher score indicates greater (i.e., "worse") interference.
Time Frame: Baseline to up to 2 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Acolbifene Hydrochloride)
Number analyzed (Participants) | 25
Participants
  Increase in HAQ score | 1
  No Change in HAQ score | 24
  Decrease in HAQ score | 0

ADVERSE EVENTS:
Time Frame: From first administration of study agent, through 2 weeks following the planned 6 month duration of study agent.
Arm/Group | Prevention (Acolbifene Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 20/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevention (Acolbifene Hydrochloride) (N=25)
Abnormal PAP smear (Reproductive system and breast disorders) | 2 (2)
Amenorrhea (Reproductive system and breast disorders) | 4 (4)
Bilateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Cervical laceration (Reproductive system and breast disorders) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased libido (Reproductive system and breast disorders) | 1 (1)
Diaphoresis (General disorders) | 1 (2) — At night 3 days during menses
Diarrhea (Gastrointestinal disorders) | 3 (5)
Finger joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Heavy bleeding with menses (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot Flashes (Endocrine disorders) | 5 (7)
Irregular menses (Reproductive system and breast disorders) | 3 (4)
Irregular prolonged menses (Reproductive system and breast disorders) | 1 (1)
Bilateral ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg cramps (Musculoskeletal and connective tissue disorders) | 3 (4)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) — Great right toe
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
Night Sweats (Endocrine disorders) | 1 (1)
Intercourse pain (Reproductive system and breast disorders) | 1 (1)
Right ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Palpable right breast mass (Skin and subcutaneous tissue disorders) | 1 (1)
Acne (scalp and neck) (Skin and subcutaneous tissue disorders) | 1 (1)
Severe mood swings (Nervous system disorders) | 1 (1)
Shingles (left flank) (Infections and infestations) | 1 (1)
Sinus infection (Infections and infestations) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stiffness in left foot (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Viral sinusitis (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Secondary to GERD
Worsening Fatigue (General disorders) | 1 (1)
Cold or allergies (Immune system disorders) | 1 (1)
Cold sores (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Intermittent diarrhea (Gastrointestinal disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes